CLINICAL TRIAL: NCT04886193
Title: Docetaxel, Oxaliplatin, Fluorouracil (FLOT Regimen) Combined With Teriprizumab (PD-1) in the First-line Treatment of Patients With Advanced Gastric Cancer and Peritoneal Metastasis: an Open, One-arm, Exploratory Study
Brief Title: FLOT Combined With PD-1 in the First-line Treatment of Patients With Advanced Gastric Cancer and Peritoneal Metastasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Collaborators: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Principal Investigator, Wei Wang, M.D., Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GDPHCM-GI-04
Record Dates: First submitted 2021-05-10; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Chemotherapy; Gastric Cancer
Keywords: FLOT, PD-1, Gastric cancer, Peritoneal metastasis
MeSH Terms: conditions — Stomach Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — S 1 (combination)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FLOT combined with PD-1 (Experimental): The enrolled patients will receive 4 cycles of FLOT regimen + teriprizumab treatment before surgery Q2W.
  If the transformation is successful, the patient undergoes R0 surgical resection of D2 lymph node dissection, and will continue to receive 4 cycles of FLOT regimen + Teripril after surgery. Anti-treatment, the treatment plan is the same as before.
  After completing the 4 cycles of treatment, oral Tiggio Capsule (S-1) and Teriprizumab were maintained for 1 year.
  Interventions: Drug: FLOT(Docetaxel+oxaliplatin+leucovorin+5-FU), Treprizumab, Tiggio capsule (S-1)

INTERVENTIONS:
Drug: FLOT(Docetaxel+oxaliplatin+leucovorin+5-FU), Treprizumab, Tiggio capsule (S-1) — * FLOT: Docetaxel 50mg/m2 ivd d1 + oxaliplatin 85mg/m2 ivd d1 + leucovorin 200mg/m2 ivd d1 + 5-FU 2600mg/m2 civ 24h Q2W
  * Treprizumab 3mg/kg, intravenously administered on the first day of each cycle, Q2W
  * Tiggio capsule (S-1) 40-60mg (BSA<1.25 m2: 40mg, 1.25 m2≤BSA≤1.5 m2: 50mg, BSA> 1.5 m2: 60mg) po bid d1-14 Q3W, continuous treatment for 1 year;
  * Teriprizumab 240mg, intravenously, given on the first day of each cycle, Q3W, continuous treatment for 1 year.

SUMMARY:
In this study, patients with advanced gastric adenocarcinoma whose peritoneal metastasis and peritoneal nodule pathologically confirmed metastasis and/or exfoliative cytology were confirmed as the clinical stage of peritoneal metastasis, who had not received treatment before, were invited to participate in the study.To evaluate the surgical conversion rate and tumor regression grade (TRG grade) of patients with stage gastric cancer with peritoneal metastasis using docetaxel, oxaliplatin, fluorouracil (FLOT regimen) combined with teriprizumab (PD-1).

DETAILED DESCRIPTION:
The study drugs in this study are docetaxel, oxaliplatin, 5-FU, leucovorin, tigio capsules and teriprizumab.

Dosage and dosing regimen for all research phases:

The enrolled patients will receive 4 cycles of FLOT regimen + teriprizumab treatment before surgery, and every 2 weeks is a treatment cycle (Q2W). The specific plan is as follows.

* FLOT: Docetaxel 50mg/m2 ivd d1 + oxaliplatin 85mg/m2 ivd d1 + leucovorin 200mg/m2 ivd d1 + 5-FU 2600mg/m2 civ 24h Q2W
* Treprizumab 3mg/kg, intravenously administered on the first day of each cycle, Q2W If the transformation is successful, the patient undergoes R0 surgical resection of D2 lymph node dissection for gastric cancer in accordance with the "Japanese Gastric Cancer Treatment Guidelines. Physician's Edition. 4th Edition". After the operation, the patient will continue to receive 4 cycles of FLOT treatment + Teripril Anti-treatment, the treatment plan is the same as before.

After completing the 4 cycles of treatment, oral Tiggio Capsule (S-1) and Teriprizumab were maintained for 1 year. The specific plan is as follows.

* Tiggio capsule (S-1) 40-60mg (BSA<1.25 m2: 40mg, 1.25 m2≤BSA≤1.5 m2: 50mg, BSA> 1.5 m2: 60mg) po bid d1-14 Q3W, continuous treatment for 1 year;
* Teriprizumab 240mg, intravenously, given on the first day of each cycle, Q3W, continuous treatment for 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent of the patient;
2. 18 years old <age <80 years old;
3. The primary gastric lesion was diagnosed as gastric adenocarcinoma by endoscopic biopsy histopathology (papillary adenocarcinoma pap, tubular adenocarcinoma tub, mucinous adenocarcinoma muc, signet ring cell carcinoma sig, poorly differentiated adenocarcinoma por);
4. The clinical stage of laparoscopic exploration is peritoneal metastasis, peritoneal nodule pathologically confirmed metastasis and/or exfoliated cytology test positive for advanced gastric cancer patients;
5. Preoperative ECOG [Using the ECOG scoring standard Zubrod-ECOG-WHO (ZPS, 5-point method) developed by the Eastern Cooperative Oncology Group (ECOG)] Physical State Score 0/1;
6. Preoperative anesthesia risk score sheet (ASA score sheet) I-III;

Exclusion Criteria:

1. The pathology of the peritoneal nodule confirmed no metastasis, and the exfoliated cytology test was negative;
2. Pregnant or lactating women;
3. Suffer from severe mental illness;
4. Preoperative imaging or intraoperative exploration revealed that there have been distant blood metastases in the liver, lungs, and brain;
5. A history of other malignant diseases within 5 years;
6. A history of allergies to any component of teriprizumab, docetaxel, oxaliplatin, and fluorouracil;
7. A history of continuous systemic corticosteroid therapy within 1 month;
8. Complications of gastric cancer (bleeding, perforation, obstruction) requiring emergency surgery;
9. A history of unstable angina or myocardial infarction, or a history of cerebral infarction or cerebral hemorrhage within 6 months, and a lung function test FEV1 <50% of the expected value;
10. Have received any of the following treatments:

    1. Have received anti-PD-1 or anti-PD-L1 antibody therapy in the past;
    2. Have received any investigational drug treatment within 4 weeks before using the drug for the first time;
    3. Enroll in another clinical study at the same time, unless it is an observational (non-interventional) clinical study or an interventional clinical study follow-up;
    4. Receive the last dose of anti-cancer treatment (including radiotherapy) within 4 weeks before the first use of the study drug;
    5. Those who have been vaccinated with anti-tumor vaccines or the study drugs have been vaccinated with live vaccines within 4 weeks before the first administration;
    6. Those who have undergone major surgery or trauma within 4 weeks before using the study drug for the first time.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Surgical conversion rate | 2-3 months
  defined as the proportion of patients who have undergone R0 surgical resection after multidisciplinary assessment after completing 4 courses of conversion adjuvant therapy
TRG grade | 2-3 months
  tumor regression grade

SECONDARY OUTCOMES:
PFS | 1 year
  Progression-free survival
OS | 1 year
  overall survival
the incidence and severity of adverse events | 1 year
  the incidence and severity of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Province Hospital of Chinese Medicine, the Second Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yamamoto M, Sakaguchi Y, Matsuyama A, Yoshinaga K, Tsutsui S, Ishida T. Surgery after preoperative chemotherapy for patients with unresectable advanced gastric cancer. Oncology. 2013;85(4):241-7. doi: 10.1159/000354420. Epub 2013 Oct 4. PMID 24107642
- [Background] Yonemura Y, Bandou E, Kawamura T, Endou Y, Sasaki T. Quantitative prognostic indicators of peritoneal dissemination of gastric cancer. Eur J Surg Oncol. 2006 Aug;32(6):602-6. doi: 10.1016/j.ejso.2006.03.003. Epub 2006 Apr 17. PMID 16617004
- [Background] Kitayama J, Ishigami H, Yamaguchi H, Yamashita H, Emoto S, Kaisaki S, Watanabe T. Salvage gastrectomy after intravenous and intraperitoneal paclitaxel (PTX) administration with oral S-1 for peritoneal dissemination of advanced gastric cancer with malignant ascites. Ann Surg Oncol. 2014 Feb;21(2):539-46. doi: 10.1245/s10434-013-3208-y. Epub 2013 Aug 22. PMID 23975319
- [Background] Bismuth H, Adam R. Reduction of nonresectable liver metastasis from colorectal cancer after oxaliplatin chemotherapy. Semin Oncol. 1998 Apr;25(2 Suppl 5):40-6. PMID 9609107
- [Background] Nakajima T, Ota K, Ishihara S, Oyama S, Nishi M, Ohashi Y, Yanagisawa A. Combined intensive chemotherapy and radical surgery for incurable gastric cancer. Ann Surg Oncol. 1997 Apr-May;4(3):203-8. doi: 10.1007/BF02306611. PMID 9142380
- [Background] Yamaguchi K, Yoshida K, Tanahashi T, Takahashi T, Matsuhashi N, Tanaka Y, Tanabe K, Ohdan H. The long-term survival of stage IV gastric cancer patients with conversion therapy. Gastric Cancer. 2018 Mar;21(2):315-323. doi: 10.1007/s10120-017-0738-1. Epub 2017 Jun 14. PMID 28616743
- [Background] Yoshida K, Yamaguchi K, Okumura N, Tanahashi T, Kodera Y. Is conversion therapy possible in stage IV gastric cancer: the proposal of new biological categories of classification. Gastric Cancer. 2016 Apr;19(2):329-338. doi: 10.1007/s10120-015-0575-z. Epub 2015 Dec 7. PMID 26643880
- [Background] Zurleni T, Gjoni E, Altomare M, Rausei S. Conversion surgery for gastric cancer patients: A review. World J Gastrointest Oncol. 2018 Nov 15;10(11):398-409. doi: 10.4251/wjgo.v10.i11.398. PMID 30487951
- [Background] Kang YK, Boku N, Satoh T, Ryu MH, Chao Y, Kato K, Chung HC, Chen JS, Muro K, Kang WK, Yeh KH, Yoshikawa T, Oh SC, Bai LY, Tamura T, Lee KW, Hamamoto Y, Kim JG, Chin K, Oh DY, Minashi K, Cho JY, Tsuda M, Chen LT. Nivolumab in patients with advanced gastric or gastro-oesophageal junction cancer refractory to, or intolerant of, at least two previous chemotherapy regimens (ONO-4538-12, ATTRACTION-2): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2017 Dec 2;390(10111):2461-2471. doi: 10.1016/S0140-6736(17)31827-5. Epub 2017 Oct 6. PMID 28993052
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Result] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Result] Al-Batran SE, Hofheinz RD, Pauligk C, Kopp HG, Haag GM, Luley KB, Meiler J, Homann N, Lorenzen S, Schmalenberg H, Probst S, Koenigsmann M, Egger M, Prasnikar N, Caca K, Trojan J, Martens UM, Block A, Fischbach W, Mahlberg R, Clemens M, Illerhaus G, Zirlik K, Behringer DM, Schmiegel W, Pohl M, Heike M, Ronellenfitsch U, Schuler M, Bechstein WO, Konigsrainer A, Gaiser T, Schirmacher P, Hozaeel W, Reichart A, Goetze TO, Sievert M, Jager E, Monig S, Tannapfel A. Histopathological regression after neoadjuvant docetaxel, oxaliplatin, fluorouracil, and leucovorin versus epirubicin, cisplatin, and fluorouracil or capecitabine in patients with resectable gastric or gastro-oesophageal junction adenocarcinoma (FLOT4-AIO): results from the phase 2 part of a multicentre, open-label, randomised phase 2/3 trial. Lancet Oncol. 2016 Dec;17(12):1697-1708. doi: 10.1016/S1470-2045(16)30531-9. Epub 2016 Oct 22. PMID 27776843
- [Result] Muro K, Chung HC, Shankaran V, Geva R, Catenacci D, Gupta S, Eder JP, Golan T, Le DT, Burtness B, McRee AJ, Lin CC, Pathiraja K, Lunceford J, Emancipator K, Juco J, Koshiji M, Bang YJ. Pembrolizumab for patients with PD-L1-positive advanced gastric cancer (KEYNOTE-012): a multicentre, open-label, phase 1b trial. Lancet Oncol. 2016 Jun;17(6):717-726. doi: 10.1016/S1470-2045(16)00175-3. Epub 2016 May 3. PMID 27157491
- [Result] Fuchs CS, Doi T, Jang RW, Muro K, Satoh T, Machado M, Sun W, Jalal SI, Shah MA, Metges JP, Garrido M, Golan T, Mandala M, Wainberg ZA, Catenacci DV, Ohtsu A, Shitara K, Geva R, Bleeker J, Ko AH, Ku G, Philip P, Enzinger PC, Bang YJ, Levitan D, Wang J, Rosales M, Dalal RP, Yoon HH. Safety and Efficacy of Pembrolizumab Monotherapy in Patients With Previously Treated Advanced Gastric and Gastroesophageal Junction Cancer: Phase 2 Clinical KEYNOTE-059 Trial. JAMA Oncol. 2018 May 10;4(5):e180013. doi: 10.1001/jamaoncol.2018.0013. Epub 2018 May 10. PMID 29543932